CLINICAL TRIAL: NCT06408909
Title: Evaluation of the Clinical Pharmacist's Effect in Achieving Treatment Goals in Hypothyroid Patients
Brief Title: Pharmacist Role in Thyroid Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other); Marmara University (Other)
Responsible Party: Principal Investigator, Muhammed Yunus Bektay, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pharm. Role Thyorid Disorder
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Hypothyroidism; Hyperthyroidism; Thyroid Diseases
Keywords: Hypothyroidism; Levothyroxine; Drug-Related Problem; Clinical Pharmacist; Medication Adherence
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism; Thyroid Diseases; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Group in which only observation is made by the clinical pharmacist For patients in this group, no intervention (i.e. recommendation) will be made to physicians by the clinical pharmacist. Within the intervention group, patient characteristics such as the underlying conditions, and the appropriateness of prescribed medications were evaluated for the patients who received levothyroxine treatment for thyroid diseases and met the inclusion criteria. The participant will take standard treatment. Evaluations will be recorded.
- Intervention Group (Experimental): Group to which the clinical pharmacist makes recommendations For patients in this group, intervention (i.e. recommendation) will be made to physician in charge by the clinical pharmacist. Within the intervention group, patient characteristics such as the underlying conditions, and the appropriateness of prescribed medications were evaluated for the patients who received treatment for thyroid diseases and met the inclusion criteria. Through medication reviews, evaluations were made to identify drug-related problems and provide solutions to these problems. The clinical pharmacist provided recommendations to the physicians regarding significant clinically important problems.
  Interventions: Behavioral: Clinical Pharmacist Intervention Group

INTERVENTIONS:
Behavioral: Clinical Pharmacist Intervention Group — Group to which the clinical pharmacist makes recommendations The drugs administered to patients during scheduled hospital visits will be recorded. A detailed medication review will be conducted by the clinical pharmacist. As a result of a comprehensive evaluation, recommendations were made to doctors regarding drug-related problems and were recorded.
  Other Names: Intervention Group
  Arms: Intervention Group

SUMMARY:
Hypothyroidism (HoT) treatment involves lifelong thyroxine replacement therapy and regular monitoring. The objective of this study was to assess the impact of clinical pharmacist (CP) intervention in managing drug-related problems (DRPs) on outcomes among hypothyroid patients receiving levothyroxine (LT4) therapy.

DETAILED DESCRIPTION:
The first choice in the treatment of hypothyroidism (HoT) is replacement therapy with levothyroxine (LT4). Factors other than the use of the drug are as crucial as the use of LT4 at the right time and in the right way. Drugs used by patients other than LT4, comorbidities, diet, age, and weight of the patient also affect the benefit seen from LT4 treatment.

LT4, which has a narrow therapeutic index, may cause drug-related problems (DRP) such as non-adherence to treatment, the timing of drug use, inappropriate use of the drug, inadequate therapeutic dose, duration of treatment, inadequate monitoring of treatment and potential drug-drug interactions (pDDI). In a study conducted in a hospital in India, DRP encountered during treatment with narrow therapeutic index drugs were compared with DRP encountered with other drugs. It was reported that DRPs were associated with pDDIs, adverse effects, dose overdose, dose underdose, untreated indications, inappropriate drug use, unnecessary drug use, and patient-related factors. In the study in which LT4 was also included, the rate of DRPs to narrow therapeutic index was 22%, and the rate of DRPs to other drugs was reported to be 8%. In a study documenting the interventions of pharmacists in hospitals in Germany, the interventions made between 2009 and 2012 were analyzed; LT4 was one of the ten drugs with the highest number of problems, and half of these problems were drug interactions and the inadequate therapeutic dose in patients with organ failure.

Aluminum hydroxide, bile acid secretagogues, calcium polystyrene sulphonate, sodium polystyrene sulphonate, calcium salts, iron preparations, multivitamin supplements containing iron, lanthanum carbonate, sevelamer, magnesium salts, orlistat, and raloxifene cause D-level drug interactions with LT4. In the concomitant use of calcium salts with LT4, it is observed that LT4 absorption and, consequently, therapeutic effect decreases [8,9]. In a systematic review of the concomitant use of LT4 and proton pump inhibitors (PPI) in hypothyroid patients with dyspepsia, gastroesophageal reflux, or peptic ulcer, a statistically significant increase in thyroid-stimulating hormone (TSH) levels was observed.

Since the therapeutic index of the LT4 drug is narrow, it emphasizes the importance of adherence to the drug in reaching ideal TSH levels. Medication adherence is a dynamic process closely linked to treatment outcomes in patients with chronic diseases. Very few studies exist on LT4 treatment and patient adherence to treatment. In their study, Yavuz et al. emphasized that almost half of HoT patients had serum TSH values outside the reference range despite receiving LT4 treatment and that adherence with LT4 treatment was one of the most critical determinants in reaching target TSH levels.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of Thyroid Disease (ICD-10 codes: E03.9)
2. Patients visited the endocrinology diseases outpatient clinic
3. Being 18 years or older.
4. Patients who could be evaluated by the clinical pharmacist for at least 24 hours within the intervention group.

Exclusion Criteria:

1. Being under 18 years old.
2. Lost follow up in 30th day after thyroid disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of suggested intervention (number) | From the date of randomization until there are 18 patient participants in each group. Average 6 months.
  Acceptance rate of suggested intervention. Drug-related problems and recommendations are classified according to PCNE (Pharmaceutical Care Network Europe) version 9.1. It was recorded how many suggestions were made in the intervention group and how many of these suggestions were accepted.
Serum Thyroid Stimulating Hormone Levels | From the date of randomization until there are 18 patient participants in each group. Average 6 months.
  Serum Thyroid Stimulating Hormone Levels
Having serum T4 Levels within the normal range | From the date of randomization until there are 18 patient participants in each group. Average 6 months.
  Having serum T4 Levels within the normal range
Change in medication adherence rate for patients with thyroid disorders | From the date of randomization until there are 18 patient participants in each group. Average 6 months.
  Change in medication adherence rate for patients with thyroid disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayhan YE, Bektay MY, Gogas Yavuz D, Sancar M. Evaluation of the clinical pharmacist's effect on achieving treatment goals in patients with hypothyroidism: a randomized controlled trial. BMC Endocr Disord. 2025 Apr 8;25(1):94. doi: 10.1186/s12902-025-01914-3. PMID 40200273